CLINICAL TRIAL: NCT01123876
Title: A Phase 1 Open-Label, Dose-Escalation Study of Veliparib in Combination With Bimonthly FOLFIRI in Subjects With Advanced Solid Tumors
Brief Title: Evaluating the Safety and Tolerability of the Poly-ADP Ribose (PARP) Inhibitor With FOLFIRI in Subjects With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-977
Record Dates: First submitted 2010-04-09; First posted 2010-05-14 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Veliparib and FOLFIRI (Experimental): Veliparib in combination with FOLFIRI regimen.
  Interventions: Drug: Veliparib

INTERVENTIONS:
Drug: Veliparib — Subjects will be given Veliparib twice daily on Days 1-5 and 15-19 every 28 days orally
  Other Names: ABT-888, Veliparib

SUMMARY:
Assess whether the combination of ABT-888 with FOLFIRI has activity in subjects with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subjects in the dose escalation cohorts must have: * Subjects with histologically or cytologically confirmed malignancy that is meta static or unresectable and for which standard curative measures or other therapy that may provide clinical benefit do not exist or are no longer effective or for whom treatment with FOLFIRI is a viable option.
3. Subjects in the expanded safety cohort must have: * Histological confirmed advanced colorectal cancer.
4. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1.
5. Subject must have adequate hematologic, renal and hepatic function as follows: * Bone Marrow: Absolute neutrophil count ANC >= 1,500/mm3; Platelets >= 100,000/mm3; Hemoglobin >= 9.5 g/dL; * Renal function: Serum creatinine < 1.5 * upper normal limit of institution's normal range OR creatinine clearance <= 50 mL/min/1.73m2 for subjects with creatinine levels above institutional normal; * Hepatic function: AST and ALT <= 2.5 * the upper normal limit of institution's normal range. For subjects with liver metastases, AST and ALT <= 5 * the upper normal limit of institution's normal range; * Bilirubin <= 1.5 * the upper normal limit of institution's normal range;
6. Partial Thromboplastin Time (PTT) must be <= 1.5 * the upper normal limit of institution's normal range and INR < 1.5. Subjects on anticoagulant (such as Coumadin) will have PTT and INR as determined by the investigator.
7. Women of childbearing potential must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and for 90 days following completion of therapy. Women of childbearing potential must have a negative serum pregnancy test within 21 days prior to initiation of treatment and/or post menopausal women must be amenorrheic for at least 12 months to be considered of non childbearing potential. * Total abstinence from sexual intercourse (minimum one complete menstrual cycle); * Vasectomized partner of female subjects; * Hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration; * Double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream); * IUD (Intra-Uterine Device); * Additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 90 days following completions of therapy.
8. Subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.
9. The subject has received up to 3 prior DNA damaging agents or cytotoxic chemotherapy treatments (prior therapies with biologic agents including, IL -2, interferon, vaccines, immunostimulants and signal transduction inhibitors are allowed) Chemotherapy received as adjuvant therapy before 2 years will not be considered as prior chemotherapy.

Exclusion Criteria:

1. Subject has received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, biologic or any investigational therapy within 28 days prior to study drug administration. Subjects receiving hormone therapy, bisphosphonates or LHRH-agonists are eligible. Subjects who have not recovered to within one grade level (not to exceed Grade 2) of their baseline following a significant adverse event or toxicity attributed to previously anti-cancer treatment are excluded.
2. Subjects in the expanded safety cohorts only, have previously been treated with a PARP inhibitor.
3. Subjects with a known history of brain metastases and primary CNS tumors
4. Subjects with a known hypersensitivity to CPT11, 5-FU or Folinic Acid.
5. Clinically significant and uncontrolled major medical condition(s) including but not limited to: * Uncontrolled nausea/vomiting/diarrhea; * Active uncontrolled infection; * Symptomatic congestive heart failure; * Unstable angina pectoris or cardiac arrhythmia; * Psychiatric illness/social situation that would limit compliance with study requirements. * Gilbert's Syndrome * Any medical condition, which in the opinion of the study investigator, places the patient at an unacceptably high risk for toxicities
6. Subjects that are being treated with Ketoconazole, enzyme-inducing anticonvulsants, and or St. John's Wort.
7. Subject is pregnant or lactating.
8. Subject who requires parenteral nutrition, tube feeding or has evidence of partial bowel obstruction or perforation within 28 days prior to study drug administration.
9. The subject has had another active malignancy within the past 3 years except for any cancer in situ that the Principal Investigator considers to be cured.
10. Previous exposure to Irinotecan.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Determine the MTD and establish the recommended phase 2 dose of Veliparib in combination with two different FOLFIRI regimens that include a reduced regimen (150 mg/m2 irinotecan) and the standard regimen (180 mg/m2) in subjects with advanced solid tumors | Screening to follow up visit

SECONDARY OUTCOMES:
To assess the safety and tolerability, pharmacokinetic profile of the combination at each of the FOLFIRI regimens. | Screening to follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Shepherd, MD, Study Director — AbbVie
Locations (8):
- United States (6):
  - Site Reference ID/Investigator# 24987, Scottsdale, Arizona
  - Site Reference ID/Investigator# 24985, Los Angeles, California
  - Site Reference ID/Investigator# 26742, Los Angeles, California
  - Site Reference ID/Investigator# 24986, Washington D.C., District of Columbia
  - Site Reference ID/Investigator# 24922, Durham, North Carolina
  - Site Reference ID/Investigator# 24983, Nashville, Tennessee
- South Korea (2):
  - Site Reference ID/Investigator# 75713, Seoul
  - Site Reference ID/Investigator# 75714, Seoul

REFERENCES:
- [Background] Jou E, Rajdev L. Current and emerging therapies in unresectable and recurrent gastric cancer. World J Gastroenterol. 2016 May 28;22(20):4812-23. doi: 10.3748/wjg.v22.i20.4812. PMID 27239108
- [Background] Berlin J, Ramanathan RK, Strickler JH, Subramaniam DS, Marshall J, Kang YK, Hetman R, Dudley MW, Zeng J, Nickner C, Xiong H, Komarnitsky P, Shepherd SP, Hurwitz H, Lenz HJ. A phase 1 dose-escalation study of veliparib with bimonthly FOLFIRI in patients with advanced solid tumours. Br J Cancer. 2018 Apr;118(7):938-946. doi: 10.1038/s41416-018-0003-3. Epub 2018 Mar 12. PMID 29527010